CLINICAL TRIAL: NCT05390541
Title: Increasing HIV/STI Home Testing, Linkage to Care, and Linkage to PrEP Via a Digital Intervention Among Black Women in a Geographic Hotspot
Brief Title: Increasing HIV/STI Home Testing Via a Digital Intervention Among Black Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00023755; 7R34MH128054-03 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-25 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hiv; Sexually Transmitted Diseases; Economic Problems
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the intervention or educational control conditions. Participants in both conditions will receive HIV/STI self-testing kits. The intervention condition will have 5 tailored sessions over 4 weeks. The education control condition will have 5 generic sessions equally dispersed over 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Control (Active Comparator): Participants will receive a generic standard of care via a combination of videos, audio, and text/graphics across 5 sessions during 4 weeks.
  Interventions: Other: Educational Control
- Empowered to Test Yourself (Experimental): There will be 5 tailored web based sessions of the intervention over 4 weeks, all of which will follow the same format.
  Interventions: Behavioral: Empowered to Test Yourself

INTERVENTIONS:
Behavioral: Empowered to Test Yourself — There will be 5 sessions of the intervention, all of which will follow the same format. Participants will be sent push notifications for each session. Each session will begin with using relevant constructs from sIMB (i.e., information and behavioral skills). Next, participants will choose positive outcomes resulting from the behavior, barriers to performing the behavior (mental contrasting), select situational cues and action plans to overcome selected barriers (implementation intentions), and practice typing in implementation intentions and positive outcomes from memory (memory practice). To ensure participants retain the implementation intentions, the investigators will use memory practice. Participants will be asked to self-code if the participant is correct or incorrect. Lastly, participants will learn behavioral skills to engage in each of the 5 actions to increase self-efficacy.
  Arms: Empowered to Test Yourself
Other: Educational Control — Participants will receive the HIV/STI home testing kit, instructions to mail in the kit, notification when results are ready to check online, treatment from a provider at Kind Clinic for positive results, and referral to Kind Clinic for PrEP. Each session and assessment will occur every 3 days. Session 1: Basic information about STIs. Session 2: HIV and stigma, basic information about HIV, and HIV transmission facts and myths. Session 3: Four stories about different people who are HIV-positive, how HIV was contracted, and one story about a woman who contracted herpes and how to all cope and live healthy lives. Session 4: How to disclose positive STI status. Session 5: Basic information about PrEP, and information on how to correctly use a male condom, female condom, and dental dam.
  Arms: Educational Control

SUMMARY:
The proposed intervention is a web-based intervention guided by theoretical components to increase HIV home testing among Black women at risk for HIV and sexually transmitted infections (STIs) in a HIV hotspot in the South. The intervention will promote using the home test, linkage to care, and linkage to pre-exposure prophylaxis (PrEP) evaluation. The intervention has the potential to be implemented on a large scale and tailored based on location and population to increase testing, treatment, and PrEP adoption.

DETAILED DESCRIPTION:
In Travis County, Texas, deemed a HIV geographic hotspot due to high HIV rates, Black women are 18.4 times more likely to contract HIV compared to women of other races/ethnicities. Black women also have higher rates of sexually transmitted infections (STIs) than other women; many STIs have no symptoms, are undiagnosed, and are untreated. Having an STI triples one's risk for contracting HIV. In Travis County, over 20% of women learned one year after contracting HIV that the the individual is HIV-positive, highlighting barriers to testing. Home HIV/STI testing has promise to increase rates of testing by circumventing barriers and thereby reduce medical costs through early detection and care. Home HIV/STI testing is also a prime opportunity to link Black women at high risk for HIV to pre-exposure prophylaxis (PrEP). Yet, home testing alone may not overcome all barriers. Pairing home testing with an intervention designed to increase motivation and overcome barriers has the most promise to increase HIV/STI testing rates. The proposed project draws on 3 components, the situated, information-motivation-behavioral (sIMB) model, mental contrasting, and implementation intentions to develop a new, web-based intervention. This intervention is comprised of 5 sessions: 1) using the HIV/STI home testing kit, 2) mailing in the kit, 3) checking results, 4) obtaining treatment, and 5) attending an appointment for PrEP. Each session is structured the same: information regarding the importance of each behavior (i.e., taking the home test, mailing in the test, checking results, linkage to care, and linkage to PrEP), motivation via mental contrasting (identifying positive outcomes and barriers to each session) and methods to overcome the identified barriers (implementation intentions), and behavioral skills to increase self-efficacy. The project will occur in 3 phases that coincide with the aims to develop and culturally tailor the intervention. 1) Conduct formative research to develop the intervention. Four focus groups (n=4-6), with 24 Black women from Travis County will explore the constructs of sIMB, mental contrasting, and implementation intentions to develop the intervention protocol to be field tested in Aim 2. 2) Field test the intervention. The investigators will test the preliminary feasibility and acceptability of the intervention with 6 participants to make any necessary adjustments for Aim 3. 3) Conduct a feasibility pilot of the intervention. The investigators will determine the feasibility, acceptability, and preliminary efficacy among 60 Black women in Travis County. Participants will be randomly assigned to the intervention or a web-based educational control. The investigators hypothesize that the intervention will be feasible, acceptable, and demonstrate a trend toward efficacy for completion of home testing, linkage to care, and linkage to PrEP. Follow-up web-based assessments will be administered 2-, 4-, and 6-months after baseline. The web-based design of the intervention greatly increases the opportunity for implementation on a large scale. The long-term goal is to increase HIV/STI testing among low-income Black women via scalable and sustainable methods to decrease HIV transmission and subsequent disparities.

ELIGIBILITY:
Inclusion Criteria:

* 15 - 59 years of age
* Identify as a cisgender woman
* Identify as Black/African-American (Black/African American mixed race/ethnicity is included)
* Read/speak/type in English
* Have not tested for HIV/STIs in the past 12 months
* Live in urban or suburban areas in Austin, Dallas, Houston, or San Antonio, Texas
* Had condom-less sex in the past 6 months
* Have access to a device (i.e., smart phone, tablet, or computer/laptop)
* Have access to the internet
* Reports at least one of the following:
* A sexual partner who is living with HIV
* Does not use or uses condoms inconsistently for vaginal/anal sex
* Injects drugs with a partner who is living with HIV
* Shared drug preparation or injection equipment with others

Exclusion Criteria:

* Over the age of 59 or younger than 15 years
* Identify as any gender other than a cisgender woman
* Identify as any race/ethnicity other than Black/African-American
* Are unable to fluently speak, read, or type in English
* Had an HIV/STI test within the past 12 months
* Live in rural areas of Texas or urban/suburban areas other than Austin, Dallas, Houston, or San Antonio, Texas
* Use condoms 100% of the time during vaginal/anal sex in the past 6 months
* Do not have access to a device (i.e., smart phone, tablet, or computer/laptop)
* Do not have access to the internet
* Reports that they do not have a sexual partner who is living with HIV, always uses condoms for vaginal/anal sex, does not inject drugs with a partner living with HIV, and does not share drug preparation or injection equipment with others.

Ages: 15 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender Black women are eligible for this study.
Enrollment: 3 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who used Home HIV Test | 4 days
  Self-report of use of HIV test within 4 days of receiving the test.
Number of participants who mailed HIV test | 2 days
  Self-report of mailing at-home HIV test within 2 days; verification from Kind Clinic that test was received.
Number of participants who checked HIV results | 7 days
  Self-report of HIV test results checked within 7 days after Kind Clinic receives the at home HIV test; results verified by Kind Clinic.
Number of HIV positive participants who received HIV treatment | 7 days
  If HIV test is positive, self-report of treatment for HIV; results verified by Kind Clinic.
Number of HIV negative participants who attended PrEP evaluation | 7 days
  If HIV test is negative, self-report of attending appointment for PrEP evaluation within 7 days after receipt of negative HIV test; appointment attendance verified by Kind Clinic.

SECONDARY OUTCOMES:
Number of participants who used home STI test | 4 days
  Self-report of use of STI test within 4 days of receiving STI home test.
Number of Participants Who Received STI treatment | Within 7 days of positive HIV test
  If applicable (if STI test is positive), self-report of treatment for STI(s); results verified by Kind Clinic.
Feasibility of Intervention Measure (FIM) score | Post intervention up to 1 week
  Scale is Completely disagree (1) to Completely agree (5). Scores average 4 items; higher scores indicate greater feasibility.
Acceptability of Intervention Measure (AIM) score | Post intervention up to 1 week
  Scale is Completely disagree (1) to Completely agree (5). Scores average 4 items; higher scores indicate greater acceptability.

OTHER OUTCOMES:
Recruitment Materials Acceptability Developed by Study Team | Baseline
  Measures adapted from the Acceptability of Intervention Measure (AIM). Scale is Completely disagree (1) to Completely agree (5). Scores average 4 items; higher scores indicate greater acceptability.
Acceptability of Measures Developed by Study Team | Post intervention up to 1 week
  Measures are adapted from other researchers: 1) The questions were easy to understand. 2) The questions were respectful. 3) The intervention instructions were bothersome (reverse score). Scale is Completely disagree (1) to Completely agree (5). Scores average 3 items; higher scores indicate greater acceptability.
Acceptability of Program Instructions Developed by Study Team | Post intervention up to 1 week
  Measures are adapted from other researchers: 1) The intervention instructions were easy to understand. 2) The intervention instructions were respectful. 3) The intervention instructions were bothersome (reverse score). Scale is Completely disagree (1) to Completely agree (5). Scores average 3 items; higher scores indicate greater acceptability.
Participant Retention Rate of Intervention and Educational Control Session. | 28 days
  The proportion of participants who completed the intervention divided by how many participants started the intervention compared to the proportion of participants who completed the educational control condition divided by how many participants started the educational control condition. Larger proportions indicate higher retention rates.
Baseline demographic characteristics | Baseline
  Race, age, gender, fluent in English, location (county), smart phone and/or internet access, income, employment, insurance.
Number of participants with high sexual risk | Baseline
  Tested for HIV/STIs and unprotected sex. Testing will be measured with 3 items by asking participants have they ever been tested for each HIV/STI individually and the answer options will be 3, 6, 12, more than 12 months ago, and never. Those who responded that they had been tested will be asked what the results the results of the test (negative, positive, or they do not know). Participants who tested more than 12 months ago or never will be eligible. Unprotected sex will as if participants had unprotected vaginal or anal sex with a man in the past 12 months. Only participants who respond "yes" will be eligible.

CONTACTS AND LOCATIONS:
Overall Officials: Liesl A Nydegger, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (4):
- United States (4):
  - Johns Hopkins Bloomberg School of Public Health, Austin, Texas
  - Johns Hopkins Bloomberg School of Public Health, Dallas, Texas
  - Johns Hopkins Bloomberg School of Public Health, Houston, Texas
  - Johns Hopkins Bloomberg School of Public Health, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the findings through presentations at national and international conferences. They will also seek to publish findings in key scientific outlets. The investigators will assure that they are in compliance with NIH requirements to deposit peer reviewed publications with the PubMed Central repository, thus facilitating dissemination of findings to the scientific community and general public. The investigators will willingly share the data with scholars wishing to collaborate on publications related to the project. To improve the ease of collaboration the investigators will thoroughly document all decisions regarding how they classify and code our transcribed and quantitative data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available in the Texas Data repository within 1 year after study completion where it will remain for 5 years.

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Ondersma SJ, Chase SK, Svikis DS, Schuster CR. Computer-based brief motivational intervention for perinatal drug use. J Subst Abuse Treat. 2005 Jun;28(4):305-12. doi: 10.1016/j.jsat.2005.02.004. PMID 15925264